CLINICAL TRIAL: NCT01326806
Title: Reducing Teen Sexual Behavior: A Clinic-Based Approach
Brief Title: A Parent-Based Intervention to Reduce Sexual Risk Behavior in Adolescents
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: New York University (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: NIH_066159; R01HD066159 (NIH)
Record Dates: First submitted 2011-03-28; First posted 2011-03-31 (Estimated); Last update posted 2022-10-27 (Actual); Status verified 2019-04

CONDITIONS: Behavior and Behavior Mechanisms
Keywords: Parent-based intervention; Sexual risk behavior; Adolescents
MeSH Terms: conditions — Behavior | interventions — Nutritional Status

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Sex Education + Standard Care (Experimental): Participating mothers will receive sex education information while their child is having a physical exam.
  Interventions: Behavioral: Families Talking Together
- Hygiene & Nutrition Education + Standard Care (Active Comparator): Participating mothers will receive information on hygiene and nutrition while their child is having a physical exam.
  Interventions: Behavioral: Active Control on Hygiene & Nutrition
- No Education + Standard Care (No Intervention): Participating mothers who are passive controls will not receive any additional information while their child is having a physical exam.

INTERVENTIONS:
Behavioral: Families Talking Together — The intervention will take place in a pediatric health care clinic and will be coordinated through provider extenders when healthcare providers see youth fora non-acute care visit. A mother of the adolescent will meet with a provider extender for approximately 30 minutes while her child is being examined by a healthcare provider. During this time, the intervention will be delivered to the mother. At the conclusion of the session, the mother will be given reference materials to take home and tasks to perform to facilitate discussions about sex with her adolescent. The healthcare provider will endorse the intervention separately for mothers and adolescents. There will be one follow-up booster session administered through phone calls to increase completion probabilities of the tasks. The target behavior is sexual activity in adolescents.
  Arms: Sex Education + Standard Care
Behavioral: Active Control on Hygiene & Nutrition — The active control group will take place in a pediatric health care clinic and will be coordinated through provider extenders when healthcare providers see youth for a non-acute care visit. The mother of the adolescent will meet with a provider extender for approximately 30 minutes while her child is being examined by a healthcare provider. During this time, the active control on hygiene and nutrition will be delivered to the mother.
  Arms: Hygiene & Nutrition Education + Standard Care

SUMMARY:
The purpose of this study is to test the feasibility and efficacy of a triadic intervention designed to target both healthcare providers and parents in order to prevent adolescent sexual risk behavior in Latino and African American adolescents. The intervention will be administered in the context of mothers waiting for their children to complete a non-acute care visit.

DETAILED DESCRIPTION:
In the United States, racial and ethnic minorities suffer disproportionately from preventable diseases and conditions. Many of these problems result from health-related behaviors that are established during childhood and adolescence. Latino and African-American adolescents are at considerable risk for the negative consequences of early, risky sexual activity. This study will focus on Latino and African-American early adolescents ages 11 to 14.

The primary aim for this study will be to test and refine a triadic intervention developed for healthcare providers and parents to address the issue of sexual risk behavior among African American and Latino adolescents.

The triadic intervention will take place in a pediatric health care clinic when mothers accompany their children for a non-acute care visit. Mothers will meet with a provider extender (medical assistant, social worker, counselor) for approximately 30 minutes while their children are being examined by a healthcare provider. During this time, mothers will receive information about the problem of premature adolescent sexual activity, support in preventing or reducing their children's sexual risk behavior, instruction about how to talk with their children about sexual risk behavior, and targeted homework activities. The healthcare provider will endorse the intervention separately for mothers and adolescents. All parents will also receive one follow-up phone call to increase the probability that the homework tasks will be completed.

Participants in this study will also be assigned to one of the following three groups: an experimental group; an active control group; or a passive control group. Participants in all groups will complete three questionnaires over the course of the study to assess outcomes. Participants in the experimental and active control groups will partake in an intervention session with a provider extender. Parents in the experimental group will meet with the provider extender to discuss effective parent-adolescent communication strategies. They will also receive take-home materials to help them communicate with and parent their adolescents to reduce sexual risk behavior. Parents in the active control group will meet with the provider extender to discuss adolescent nutrition and receive informational brochures.

One booster session will take place via telephone for parents in the experimental and active control groups. The booster call will occur approximately 1 month after study entry. No such booster calls will be provided to parents in the passive control condition.

ELIGIBILITY:
Inclusion Criteria:

* Adolescents must be between the ages of 11 and 14 years old
* Adolescent is able to agree to being a participant
* Participant must be able to participate in questionnaire and intervention activities
* Participant must be of Latino or African American descent

Exclusion Criteria:

* Any cognitive or psychiatric disability that would prevent successful participation in questionnaire or intervention activities

Ages: 11 Years to 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 1800 (Actual)
Dates: Start 2012-02-15 (Actual); Primary Completion 2016-05-31 (Actual); Study Completion 2016-05-31 (Actual)

PRIMARY OUTCOMES:
Incidence of vaginal intercourse | Measured at 12 months post-intervention
Incidence of condom use | Measured at 12-months post-intervention

SECONDARY OUTCOMES:
Number of sexual partners | Measured at 12 months post-intervention
Behavioral intentions | Measured at 12 months post-intervention
  Behavioral intentions to engage in sexual intercourse will be assessed based on responses to three statements, each using a five point agree-disagree scale. The items are: (a) I think I am ready to have sexual intercourse; (b) I would have sexual intercourse now if I had a boy who would do it with me; and (c) I plan on having sexual intercourse in the next six months.
Incidence of vaginal intercourse | Measured at 3 months post-intervention
Incidence of condom use | Measured at 3 months post-intervention
Number of sexual partners | Measured at 3 months post-intervention
Behavioral intentions | Measured at 3 months post-intervention
  Behavioral intentions to engage in sexual intercourse will be assessed based on responses to three statements, each using a five point agree-disagree scale. The items are: (a) I think I am ready to have sexual intercourse; (b) I would have sexual intercourse now if I had a boy who would do it with me; and (c) I plan on having sexual intercourse in the next six months.

CONTACTS AND LOCATIONS:
Overall Officials: Vincent Guilamo-Ramos, PhD, ANP-BC, Principal Investigator — New York University
Locations (1):
- New York University, New York, New York, United States

REFERENCES:
- [Derived] Guilamo-Ramos V, Benzekri A, Thimm-Kaiser M, Dittus P, Ruiz Y, Cleland CM, McCoy W. A Triadic Intervention for Adolescent Sexual Health: A Randomized Clinical Trial. Pediatrics. 2020 May;145(5):e20192808. doi: 10.1542/peds.2019-2808. PMID 32345685